CLINICAL TRIAL: NCT05356910
Title: Onboarding Positives and PrEP Users to Engage Negatives (OPPEN): Peer-driven Education to Link YMSM of Color to PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Heather Pines, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R34MH121234 (NIH)
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPPEN Intervention (Experimental): OPPEN consists of three small-group and two one-on-one sessions to train YMSM of color engaged in HIV or PrEP care to be peer PrEP educators within their social networks.
  Interventions: Behavioral: OPPEN
- Control Condition (Other): The time- and attention-matched control condition consists of three small-group and two one-on-one sessions to support diet and nutrition behavior change.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: OPPEN — OPPEN training sessions (three small-group and two one-on-one sessions) build skills for effective peer PrEP outreach through didactic instruction, group discussions, role-play exercises, and goal planning and problem-solving activities.
  Arms: OPPEN Intervention
Behavioral: Control Condition — Control sessions (three small-group and two one-on-one sessions) build skills for diet and nutrition behavior change through didactic instruction, group discussions, and goal planning and problem-solving activities.
  Arms: Control Condition

SUMMARY:
Onboarding Positives and PrEP users to Engage Negatives (OPPEN) is an intervention to train young men who have sex with men (YMSM) of color living with HIV or using pre-exposure prophylaxis (PrEP) to promote PrEP use among HIV-negative YMSM of color in their social networks. This pilot randomized controlled trial will evaluate OPPEN's acceptability, feasibility, and preliminary effect on PrEP care engagement among YMSM of color.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis (PrEP) uptake has been slow among young men who have sex with men (YMSM), particularly those of color who experience a high rate of new HIV infections in the United States. Limited PrEP knowledge, unfamiliarity with how to access PrEP, medical mistrust, and stigma are barriers to PrEP care engagement among YMSM, including those of color. Peer-driven social network interventions that train individuals as peer educators to disseminate information about HIV prevention and treatment within their social networks have been implemented to address similar barriers and improve HIV outcomes within hard to reach populations. YMSM of color engaged in HIV/PrEP care often employ resilience processes to overcome socio-structural barriers to HIV prevention and care. As such, training YMSM of color engaged in HIV/PrEP care as peer PrEP educators may position them as credible sources of PrEP information who can influence behavior change (i.e., PrEP care engagement) among YMSM peers of color in their social networks via their ability to disseminate culturally competent PrEP messages in the context of their personal experiences using these resilience processes to navigate the healthcare system, medical mistrust, and stigma. Drawing on existing peer-driven social network interventions, the diffusion of innovations and information-motivation-behavioral skills models, and Harper et al.'s resilience framework, this study will develop and pilot Onboarding Positives and PrEP users to Engage Negatives (OPPEN), a peer-driven PrEP education social network intervention, among YMSM of color in San Diego, California. Through three small-group and two one-on-one sessions, OPPEN will train YMSM of color engaged in HIV/PrEP care to be peer PrEP educators within their social networks. In Phase I, OPPEN was developed, pretested, and refined using an iterative process that integrated feedback elicited from YMSM of color living with HIV and YMSM using PrEP trained via OPPEN as well as HIV-negative YMSM who could benefit from PrEP (AIM 1). In Phase II, OPPEN will be piloted in a randomized controlled trial with 70 YMSM of color engaged in HIV/PrEP care (i.e., indexes; up to two-thirds engaged in PrEP care) randomly assigned to OPPEN (n=35) or a time- and attention-matched control condition (n=35). All indexes will receive coupons to recruit YMSM peers of color within their social networks to the study. Assuming ~2 peers will be recruited per index, ~140 peers will present at the study site (i.e., peer-recruits) and undergo HIV testing. HIV-negative peer-recruits interested in PrEP will be scheduled for a PrEP clinic visit. Data collected via surveys (baseline and 3-month study visits) and medical records will be used to evaluate the preliminary effect of OPPEN on PrEP interest, linkage, and uptake among peer-recruits (AIM 2) and theory-based mechanisms targeted by OPPEN among indexes and peer-recruits (AIM 3). OPPEN acceptability and feasibility will be evaluated using a mixed-methods approach (AIM 4).

ELIGIBILITY:
Inclusion Criteria (Index Participants):

* 18-34 years-old
* Cisgender male
* Fluent in English
* Person of color
* Engaged in HIV care or PrEP care
* Sexual activity with cisgender men or transgender women in their lifetime
* Social networks with at least three 18-34 year-old MSM peers of color
* Willing to disclose their HIV status or PrEP use to their 18-34 year-old MSM peers of color
* Willing to provide written informed consent

Inclusion Criteria (Peer-Recruit Participants):

* 18-34 years-old
* Cisgender male
* Fluent in English or Spanish
* Person of color
* HIV-negative
* Not using PrEP
* Sexual activity with cisgender men or transgender women in their lifetime
* Willing to provide written informed consent

Exclusion Criteria:

* Persons who meet the criteria above will be eligible, no other exclusion criteria will apply.

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Persons screened for eligibility will be asked their gender identity. Those who identify as cisgender men will be eligible.
Enrollment: 78 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Pines, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon review of written requests from researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Approximately 6 months after the publication of the study's primary findings.
Access Criteria: Requests from researchers for de-identified data will be reviewed by the research team (Principal Investigator and Co-Investigators).

RESULTS

PARTICIPANT FLOW:
Groups:
- OPPEN Index Participants: Index participants randomized to receive the OPPEN intervention, which trains young men who have sex with men (YMSM) of color engaged in HIV or pre-exposure prophylaxis (PrEP) care to be peer PrEP educators within their social networks. OPPEN training sessions (three small-group and two one-on-one sessions) build skills for effective peer PrEP outreach through didactic instruction, group discussions, role-play exercises, and goal planning and problem-solving activities.
- Control Index Participants: Index participants randomized to receive the time- and attention-matched control condition, which supports diet and nutrition behavior change. Control sessions (three small-group and two one-on-one sessions) build skills for diet and nutrition behavior change through didactic instruction, group discussions, and goal planning and problem-solving activities.
- OPPEN Peer-Recruit Participants: Peers recruited to participate in the study by index participants randomized to the OPPEN intervention.
- Control Peer-Recruit Participants: Peers recruited to participate in the study by index participants randomized to the control condition.
Period: Overall Study
Arm/Group | OPPEN Index Participants | Control Index Participants | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Started | 35 | 35 | 2 | 6
Completed | 21 | 14 | 2 | 6
Not Completed | 14 | 21 | 0 | 0
Not completed — Lost to Follow-up | 10 | 19 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OPPEN Index Participants: Index participants randomized to receive the OPPEN intervention, which trains YMSM of color engaged in HIV or PrEP care to be peer PrEP educators within their social networks. OPPEN training sessions (three small-group and two one-on-one sessions) build skills for effective peer PrEP outreach through didactic instruction, group discussions, role-play exercises, and goal planning and problem-solving activities.
- Total: Total of all reporting groups
Arm/Group | OPPEN Index Participants | Control Index Participants | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants | Total
Number analyzed (Participants) | 35 | 35 | 2 | 6 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (3.5) | 26.9 (4.3) | 24.0 (1.4) | 24.0 (3.0) | 26.8 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 35 | 35 | 2 | 6 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 28 | 1 | 6 | 61
  Not Hispanic or Latino | 9 | 7 | 1 | 0 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 9 | 7 | 1 | 1 | 18
  White | 8 | 12 | 0 | 1 | 21
  More than one race | 7 | 2 | 1 | 2 | 12
  Unknown or Not Reported | 10 | 13 | 0 | 2 | 25
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 2 | 6 | 78
HIV/PrEP care engagement [Count of Participants; unit: Participants]
  Engaged in HIV care | 11 | 12 | 0 | 0 | 23
  Engaged in PrEP care | 24 | 23 | 0 | 0 | 47
  Not engaged in care | 0 | 0 | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: PrEP Interest (Peer-Recruit Participants)
Description: Participants used 5-point Likert scale responses (very uninterested to very interested) to indicate their interest in taking oral PrEP ("How interested are you in taking oral PrEP to prevent HIV?") and injectable PrEP ("How interested are you in taking injectable PrEP to prevent HIV?"). Responses of "interested" or "very interested" in either oral or injectable PrEP defined PrEP interest.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 6
Participants | 2 | 3

2. Primary Outcome: PrEP Linkage (Peer-Recruit Participants)
Description: Attended a PrEP care visit since baseline.
Time Frame: 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 6
Participants | 1 | 2

3. Primary Outcome: PrEP Uptake (Peer-Recruit Participants)
Description: Started using oral or injectable PrEP since baseline.
Time Frame: 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 6
Participants | 1 | 2

4. Secondary Outcome: PrEP Conversations With Peers (Index Participants)
Description: Reported having conversations about PrEP with at least one YMSM peer in their social network in the last three months.
Time Frame: 3-month follow-up
Population: Index participants who completed the study and reported on conversations with YMSM peers in their social networks.
Measure: Count of Participants; unit: Participants
Arm/Group | OPPEN Index Participants | Control Index Participants
Number analyzed (Participants) | 20 | 14
Participants | 15 | 9

5. Secondary Outcome: PrEP Information (Peer-Recruit Participants)
Description: Sum score on 13-item PrEP knowledge scale where higher scores indicate greater PrEP knowledge (range: 0-13).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 6
Score on a scale | 9.0 (2.8) | 5.7 (2.9)

6. Secondary Outcome: PrEP Motivation (Peer-Recruit Participants)
Description: Sum of 5-point Likert scale responses (strongly disagree to strongly agree) to scales measuring PrEP attitudes (5 items), PrEP stigma (5 items), subjective PrEP norms (6 items), and descriptive PrEP norms (6 items) where higher scores indicate greater motivation to use PrEP (range: 22-110).
Time Frame: Baseline
Population: Peer-Recruit participants who responded to all scale items.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 5
Score on a scale | 85.5 (9.2) | 77.8 (13.9)

7. Secondary Outcome: PrEP Behavioral Skills (Peer-Recruit Participants)
Description: Sum score on 8-item PrEP self-efficacy scale where higher scores indicate greater PrEP self-efficacy (range: 8-32).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 6
Score on a scale | 30.5 (0.7) | 23.5 (5.8)

8. Secondary Outcome: Session Acceptability (Index Participants)
Description: Mean score of 5-point Likert scale responses (strongly disagree to strongly agree) to 21 items measuring acceptability of OPPEN/control sessions among index participants where higher scores indicate greater acceptability (range: 1-5).
Time Frame: 3-month follow-up
Population: Index participants who completed the study and responded to all acceptability items.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OPPEN Index Participants | Control Index Participants
Number analyzed (Participants) | 17 | 14
Score on a scale | 4.5 (0.4) | 4.3 (0.4)

9. Secondary Outcome: Session Feasibility (Index Participants)
Description: Mean score of 5-point Likert scale responses (strongly disagree to strongly agree) to 5 items measuring feasibility of OPPEN/control sessions among index participants where higher scores indicate greater feasibility (range: 1-5).
Time Frame: 3-month follow-up
Population: Index participants who completed the study and responded to all feasibility items.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OPPEN Index Participants | Control Index Participants
Number analyzed (Participants) | 19 | 13
Score on a scale | 4.2 (0.7) | 3.9 (0.5)

10. Secondary Outcome: Acceptability of Interaction With Referring Index (Peer-Recruit Participants)
Description: Mean score of 5-point Likert scale responses (strongly disagree to strongly agree) to 9 items measuring the acceptability of the interaction with their peer (OPPEN or control index) when they referred them to the study among peer-recruit participants where higher scores indicate greater acceptability (range: 1-5).
Time Frame: Baseline
Population: Peer-Recruit participants who responded to all acceptability items.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 5
Score on a scale | 4.7 (0.4) | 3.6 (0.8)

11. Secondary Outcome: Feasibility of Interaction With Referring Index (Peer-Recruit Participants)
Description: Mean score of 5-point Likert scale responses (strongly disagree to strongly agree) to 2 items measuring the feasibility of the interaction with their peer (OPPEN or control index) when they referred them to the study among peer-recruit participants where higher scores indicate greater feasibility (range: 1-5).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
Number analyzed (Participants) | 2 | 6
Score on a scale | 4.5 (0.7) | 4.0 (0.6)

ADVERSE EVENTS:
Time Frame: We collected adverse event data throughout recruitment and follow-up, spanning ~2.5 years.
Arm/Group | OPPEN Index Participants | Control Index Participants | OPPEN Peer-Recruit Participants | Control Peer-Recruit Participants
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/2 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT05356910/Prot_SAP_000.pdf